CLINICAL TRIAL: NCT06883890
Title: Extended LH Administration (ELHA), a Strategy to Increase the Pool of Recruitable Antral Follicles: a Multicentric Randomized Trial
Brief Title: Extended LH Administration
Acronym: ELHA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Antonio La Marca, Professor, Azienda Ospedaliero-Universitaria di Modena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC 174/2023; 2022-004285-38 (EudraCT Number)
Record Dates: First submitted 2025-02-18; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Reserve
Keywords: AMH; AFC; Ovarian reserve; LH
MeSH Terms: interventions — Luteinizing Hormone, beta Subunit

STUDY DESIGN:
Intervention Model Description: Two-arm, multicenter, prospective, RCT (proof of concept) trial with two treatment arms at 2:1 ratio will involve couples attending an IVF/ICSI cycle, phase II study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LH group (Active Comparator): In the treatment group patients will receive the pretreatment with rLH, a daily dose of 187.5 IU (75 U in the morning and 112.5U in the evening) rLH treatment for 60 days will be administered
  Interventions: Drug: Recombinant LH (Luveris)
- Control group (Sham Comparator): In the control group, women will not receive any therapy and will be followed up with the same schedule as women in the treatment group
  Interventions: Drug: No Treatment Added

INTERVENTIONS:
Drug: Recombinant LH (Luveris) — In the treatment group patients will receive the pretreatment with rLH, a daily dose of 187.5 IU (75 U in the morning and 112.5U in the evening) rLH treatment for 60 days will be administered.
  Arms: LH group
Drug: No Treatment Added — In the control group, women will not receive any therapy and will be followed up with the same schedule as women in the treatment group
  Arms: Control group

SUMMARY:
Luteinizing hormone (LH) plays an important role in follicular development, especially in the later stages of folliculogenesis. Theca interstitial cells and, later, granulosa cells express high concentrations of receptors for LH (LH-R). LH modulates the progressive remodeling and growth of the follicle .

New evidence points to a role for LH in promoting ovarian follicle growth and maturation, even at very early stages of folliculogenesis. Studies analyzing LH-R expression profiles in the ovary have shown that LH-R is moderately expressed even in the smallest follicles, during what is known as the gonadotropin-independent phase . Immunohistochemical studies that examined the localization of LH-R in human follicles through different stages of follicular development reveal that LH-R is expressed by granulosa cells and some thecal cells in small pre-antral follicles LH promotes the transition of follicles to the antral stage, thus leading to an increase in functional ovarian reserve. Early follicular stages, particularly those between the primordial and pre-antral stages, are critical as they regulate the rate of follicle recruitment. The potential roles of LH in the early follicular phase were analyzed in a prospective, randomized multicenter study using a sequential approach to stimulation with recombinant human r-LH, followed by r-FSH, in women in hypogonadotropic hypogonadism because they were profoundly down-regulated by the administration of depo agonist GnRH analog. LH treatment was associated with an increase in small antral follicles before FSH stimulation and a higher number of normally fertilized embryos. In addition, AMH hormone was found to be significantly increased in both groups during the week prior to FSH stimulation These results seem to indicate that, if the reduction in the number of antral follicles is not due to a decrease in the number of primordial follicles, but to a slowing of progression, as in the case of women with long-standing hypothalamic amenorrhea, there may be room for a therapeutic approach. This is with the aim of improving the response to ovarian stimulation of the aforementioned patients who present with anovulatory cycles and in a condition of hypogonadotropic hypogonadism.

A recent case series described two patients suffering from hypothalamic amenorrhea with very low levels of endogenous gonadotropins, and ovulatory factor infertility. These patients were treated with exogenous LH for one to two months (prolonged administration of LH). Increased levels of both AMH and AFC were demonstrated, and they responded adequately to ovarian stimulation.

The purpose of this multicenter prospective randomized study follows recent publications confirming the implementation of ovarian reserve by supplementation with pretreatment with r-LH, a drug already on the market and routinely used in conventional controlled ovarian stimulation protocols.

The aim is to confirm that pretreatment with rhLH at a dose of 185.5 IU/day for 60 days can improve ovarian reserve, as indicated by increased baseline AMH and AFC, compared with no pretreatment. The primary outcome is serum AMH value after treatment with r-LH and without.

The planned duration of the study is 18 months, and a total of 84 patients are to be recruited. Patients will be randomized into two groups: group A who will receive pre-treatment with r-LH 185.5IU/day for 60 days and group B who will not receive pre-treatment.

Patients will have a monitoring visit every two weeks for the duration of treatment, during which an ultrasound and blood sampling will be performed to evaluate the hormonal picture. Following pretreatment, a visit of with assessment of serum AMH and AFC value will be performed and the planned IVF cycle will be started. This will be followed by an additional final follow-up visit to collect obstetric and newborn outcomes that will be conducted by telephone

DETAILED DESCRIPTION:
Primary objective The primary endpoint of the study will be to confirm that the pre-treatment with rhLH at the dose of 187.5 IU/day for 60 days may improve ovarian reserve as indicated by an increase in basal AMH.

The primary endpoint of the study will be to confirm that the pre-treatment with rhLH at the dose of 187.5 IU/day for 60 days may improve ovarian reserve as indicated by an increase in basal AMH. The chosen dose and duration for the study was based on a recent published article. In particular in this study women who presented for fertility treatment with very low functional ovarian reserve, showed that the administration of LH 187.5 IU/day for 60 days, contributed to a clinically evident increase in the functional ovarian reserve (AFC and AMH levels). The use of recombinant LH in women with gonadotrophin deficiency has been already investigated in two very well known randomized trials. In these two trials a dose of rec LH up to 225IU daily has been tested.

The objective of the European Recombinant Human LH study group was to conduct a randomized, efficacy clinical study with rLH in order to determine the minimal effective dose of rLH for supporting rFSH-induced follicular development in LH- and FSH-deficient anovulatory women (HH) in addition to assessing the safety and tolerability of this treatment. Patients were randomized to receive rLH (0, 25, 75, or 225IU/day) in addition to a fixed dose of rFSH (150 IU/day). rhLH was found 1) to promote dose-related increases in estradiol (E2) and androstenedione secretion by rFSH-induced follicles, 2) to increase ovarian sensitivity to FSH, as demonstrated by the proportion of patients who developed follicles after the administration of a fixed dose of FSH, and 3) to enhance theability of these follicles to luteinize when exposed to hCG. Recombinant LH, given sc at a dose up to 225 IU/day, was not immunogenicand was well tolerated.

In one study two double-blind, placebo-controlled, multicentre pilot studies were conducted. Study A was conducted in hypogonadotrophic hypogonadal women (WHO group I anovulation) with severe deficiency in LH and who were willing to conceive. Study B was conducted in WHO group II anovulatory patients (PCO) willing to conceive and who over-responded to FSH therapy. In the study A women received FSH plus LH at a dose of 225 IU daily. In the study B women were randomized to receive a dose of 225 IU or 450 IU daily. Authors reported that the Treatment with rLH was well tolerated. There were no serious or signficant adverse events during the study. No patient developed anti-LH antibodies.

Secondary objectives

The secondary endpoints will be:

1. Change from baseline for basal AFC (antral follicle count) after 60 days of LH prolonged treatment or no treatment
2. Change from baseline for basal AMH after 30 days of LH prolonged treatment or no treatment
3. Change from baseline for basal AFC (antral follicle count) after 30 days of LH prolonged treatment or no treatment
4. Ovarian response to controlled ovarian stimulation in IVF/ICSI cycles (number of follicles >16 mm at the end of stimulation, number of retrieved oocytes, FORT index- follicles to oocyte ratio, number of mature oocytes)
5. Evaluate the safety of rLH throughout the treatment period
6. cycles discontinued/cancelled before rhCG administration due to poor or excessive ovarian response
7. percent of missed transfer of fresh embryos
8. implantation rate
9. biochemical pregnancy rate
10. clinical pregnancy rate
11. early (≤9 days after triggering) and late (12-17 days after triggering) OHSS onset (according to Golan's Classification System) rate
12. miscarriage rate
13. preterm birth rate
14. low birth weight rate
15. congenital anomalies rate
16. gestational age at delivery
17. mean neonatal weight

This is a multicenter clinical trial. The coordinating center is the Mother-Infant Department of University Hospital of Modena and Reggio Emilia (Principal investigator [PI]: Prof. La Marca Antonio)

This two-arm, multicenter, prospective, RCT (proof of concept) trial with two treatment arms at 2:1 ratio will involve couples attending an IVF/ICSI cycle, phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. AFC of at least 5 in the 3 months prior to the study cycle
2. Basal AMH levels of at least 1 ng/ml in the 3 months prior to the study cycle
3. Age 25-38 at the moment of the study cycle
4. D3 Basal LH: 1-6 IU/L in the 3 months prior to the study cycle
5. D3 Basal FSH: < 8 IU/L in the 3 months prior to the study cycle 13
6. D3 Estradiol < 70 pg/ml in the 3 months prior to the study cycle
7. Willing to participate
8. Capable to understand and follow the study procedure
9. eumenorrheic women with low LH levels candidate to IVF/ICSI cycle for tubal factor, male factor or for idiopathic infertility
10. Acceptance and signature of the informed consent

Exclusion criteria:

1. PCOS patients according to Rotterdam's criteria
2. Patients with irregular cycles (shorter than 25 days or longer than 35 days)
3. Patients already treated with LH priming
4. Patients planning to undergo duo/double stimulation
5. Patients with ASRM Stage III or IV endometriosis
6. Patients with prior surgery significantly affecting ovary (ie ovariectomy, cystectomy significantly reducing ovarian volume or others) as assessed by the responsible gynecologist
7. Previous cycle with less than 4 oocytes recovered
8. Patients treated with hormones in the 3 months before the study
9. Patients with an already known endocrinological disease including hypothyroidism (defined by TSH < 4 mIU/L), adrenocortical deficiency (ACTH stimulation test (250 mcg) with basal cortisol <3 mcg or, if basal cortisol is 3-18 mcg serum level, cortisol serum level 30 minutes after the stimulation test <18 mcg) and hyperprolactinemia (PLR > 25mcg/l)
10. previous episode of OHSS or exuberant ovarian response to gonadotropins
11. hypersensitivity to the study drug
12. contraindication for pregnancy
13. porphyria or a family history of porphyria
14. history of ovarian torsion
15. BMI > 30 kg/m2
16. ovarian enlargement or ovarian cyst
17. gynecological bleeding of unknown origin
18. history of ovarian, breast or endometrial cancer.

Ages: 25 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Anti-Mullerian Hormone | up to 18 months
  The primary endpoint of the study will be to confirm that the pre-treatment with rhLH at the dose of 187.5 IU/day for 60 days may improve ovarian reserve as indicated by an increase in basal AMH

SECONDARY OUTCOMES:
Antral follicle count | up to 18 months
  Change from baseline for basal AFC (antral follicle count) after 60 days of LH prolonged treatment or no treatmen

CONTACTS AND LOCATIONS:
Overall Officials: Antonio La Marca, MD, PhD, Principal Investigator — University of Modena and Reggio Emilia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] La Marca A, Longo M. Extended LH administration as a strategy to increase the pool of recruitable antral follicles in hypothalamic amenorrhea: evidence from a case series. Hum Reprod. 2022 Oct 31;37(11):2655-2661. doi: 10.1093/humrep/deac195. PMID 36107111